CLINICAL TRIAL: NCT03276650
Title: Admission of Adult-onset Still Disease Patients in the ICU: a French Retrospective Multicentric Study
Brief Title: Admission of Adult-onset Still Disease Patients in the ICU
Acronym: Still-ICU
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/Still-ICU-LEMARIE/VS
Record Dates: First submitted 2017-08-25; First posted 2017-09-08 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Adult-Onset Still Disease; Critically Ill
MeSH Terms: conditions — Still's Disease, Adult-Onset; Critical Illness | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill AOSD patients: no intervention Data collection from hospitalisation reports (administrative, biological, clinical, outcome)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — biological, administrative, clinical, outcome date

SUMMARY:
Since its first description in 1971, diagnosing adult-onset Still's disease (AOSD), a rare multisystemic disorder considered as a multigenic autoinflammatory syndrome, remains challenging. Rarely, AOSD may present severe systemic manifestations and require intensive care. The main purpose of the Stil ICU study is to make the first description of the epidemiology of critically ill AOSD patients. The investigators will use a retrospective cohort study design with dual recruitment strategies: (1) via the AOSD referral centres network and (2) via a French academic medical ICU network.

ELIGIBILITY:
Inclusion Criteria:

* AOSD (history of newly diagnosed)
* ICU admission between January 2001 and June 2017

Exclusion Criteria:

* adults under protection
* admission in step-down unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AOSD patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
number of patients | At inclusion
  Number of patients fulfilling the inclusion criteria

SECONDARY OUTCOMES:
APACHE II | 24hour after ICU admission
  Acute Physiologic Assessment and Chronic Health Evaluation II
Mortality | through study completion, maximum 17,5 years after admission
  Kaplan Meier
Number of rehospitalisation in ICU | through study completion, maximum 17,5 years after admission
  need for critical care after the first hospitalisation in ICU
number of hospitalisation in internal medicine ward | through study completion, maximum 17,5 years after admission
  number of hospitalisation in internal medicine ward after the first ICU stay
recurrent relapses | through study completion, maximum 17,5 years after admission
  number of recurrent flares after the first hospitalisation in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: No